CLINICAL TRIAL: NCT04812496
Title: Tenofovir-DF Versus Hydroxychloroquine in the Treatment of Hospitalized Patients With COVID-19: An Observational Study (TEDHICOV)
Brief Title: Tenofovir-DF Versus Hydroxychloroquine in the Treatment of Hospitalized Patients With COVID-19 (TEDHICOV)
Acronym: TEDHICOV
Status: Completed | Type: Observational
Sponsor: Hospital Nacional Carlos Alberto Seguin Escobedo - EsSalud (Other)
Responsible Party: Principal Investigator, Mario Cornejo-Giraldo, Head of the Infectious Diseases Unit, Principal Investigator, Hospital Nacional Carlos Alberto Seguin Escobedo - EsSalud
Other Study IDs: TEDHICOV
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Covid19; SARS-CoV Infection; Tenofovir
Keywords: Covid-19; SARS-CoV-2; Tenofovir; Hydroxychloroquine; Hospitalized
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although several therapeutic agents have been suggested for the treatment of the disease caused by the Coronavirus of the year 2019 (COVID-19), no antiviral has yet demonstrated consistent efficacy.

This is an observational study comparing Tenofovir-DF (disoproxil fumarate) (TDF) with Hydroxychloroquine (HCQ) in the treatment of hospitalized patients with COVID-19 with evidence of pulmonary compromise and with supplemental oxygen required.

DETAILED DESCRIPTION:
All hospitalized patients with COVID-19 from March 2020 to May 30, 2020 at the "Hospital Nacional Carlos Alberto Seguín Escobedo (CASE)-EsSalud" (Arequipa, Peru) with a PCR-confirmed diagnosis of SARS-CoV-2 will be included.

The primary outcomes to be compared will be mortality, the need for admission to the Intensive Care Unit (ICU) and / or Mechanical Ventilation, and LOS (length of stay) in both groups.

Furthermore, demographic factors, risk factors, vital / respiratory functions, and laboratory results of both groups will be compared. The tests closest to the time of admission to the hospital will be taken into consideration.

Statistical Analysis: quantitative variables will be expressed as mean ± standard deviation, qualitative variables will be expressed as percentages (%). In the univariate analysis, the Student's t test will be used for the means and the chi2 test for nominal or ordinal variables. Kaplan-Meier survival curves will be evaluated 30 days after admission to the hospital to assess mortality. The multivariate analysis of the variables that result significant in the univariate analysis will be carried out by the Cox regression model in the evaluation of mortality; the multivariate linear regression model for the evaluation of the stay and the "log rank" model for the evaluation of admission to the Intensive Care Unit (ICU) or the need for mechanical ventilation (MV). In addition, models will be developed to estimate the effects of TDF treatment by regression adjustment for the primary outcomes of this observational study: hospital stay, need for ICU (intensive care unit) and / or MV (mechanical ventilation) and mortality. The Stata® software version 14 will be used and p <o.o5 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adults over 18 years of age
* Positive molecular test for SARS-CoV-2
* Computed tomography (TC scan) compatible with "COVID pneumonia" and / or in need of supplemental oxygen
* Therapy with Tenofovir-DF (TDF) or Hydroxychloroquine (HCQ) at least 3 days
* Signed informed consent

Exclusion Criteria:

* Negative molecular test for SARS-CoV-2
* No need for hospitalization
* Negative CT scan for "COVID pneumonia" and / or no supplemental oxygen requirement for COVID-19
* Had not received either HCQ or TDF, or both drugs at the same time, or had received HCQ or TDF for two days or less
* No signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients over 18 years of age hospitalized with Pneumonia COVID-19 between March and May 2020 in the Hospital Nacional CASE-EsSalud
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Mortality within 30 days of hospital admission | 30days
  Patients with COVID-19 who died within 30 days of hospitalization
Mechanical Ventilation | 30 days
  Patients with COVID-19 who required mechanic ventilation during hospitalization
Hospital stay | 30 days
  Length of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Mario Cornejo-Giraldo, M.D., Principal Investigator — Head of the Infectious Diseases Unit
Locations (1):
- Hospital Nacional CASE - EsSalud, Arequipa, Peru

IPD SHARING:
Plan to Share IPD: Yes
It is planned that all patient data included in the study will be shared after publication of the study minus those that allow the identification of the same patients
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be shared within 30 days of the publication of the study.
Access Criteria: The study data will be shared indefinitely for the benefit of the search for adequate therapy against COVID-19